CLINICAL TRIAL: NCT04114058
Title: Pain Outcomes Following Hip Arthroscopy: A Prospective Randomized Control Study Comparing Fascia Iliaca Blockade vs Extracapsular Local Field Infiltration With Liposomal Bupivacaine
Brief Title: A Study Comparing Fascia Iliaca Blockade vs Extracapsular Local Field Infiltration With Liposomal Bupivacaine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Michael Banffy, MD, Director, Orthopaedic Sports Medicine Fellowship, Cedars-Sinai Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00056482
Record Dates: First submitted 2019-09-04; First posted 2019-10-03 (Actual); Results first posted 2021-05-11 (Actual); Last update posted 2021-05-11 (Actual); Status verified 2021-04

CONDITIONS: Femoro Acetabular Impingement
Keywords: hip arthroscopy
MeSH Terms: conditions — Femoracetabular Impingement

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Liposomal Bupivicaine (Active Comparator): Following hip arthroscopy, local field infiltration with liposomal bupivicaine will be performed for adjunct pain control
  Interventions: Drug: liposomal bupivicaine
- fascia iliaca blockade (Active Comparator): Preoperatively before hip arthroscopy, a fascia iliaca blockade will be performed for adjunct pain control
  Interventions: Procedure: Fascia iliaca blockade

INTERVENTIONS:
Drug: liposomal bupivicaine — local field infiltration
  Other Names: exparel
  Arms: Liposomal Bupivicaine
Procedure: Fascia iliaca blockade — fascia iliaca compartment blockade
  Arms: fascia iliaca blockade

SUMMARY:
The purpose of this study is to compare the effectiveness of fascia iliaca blockade vs local field infiltration with liposomal bupivicaine in controlling pain, narcotic utilization and falls in the postoperative period following hip arthroscopy

DETAILED DESCRIPTION:
The purpose the research is to help determine optimal means of post-operative analgesia following hip arthroscopic procedures. Post-operative pain is a significant contributor to patient satisfaction and the side effects of narcotic pain medication are well described. The ideal intervention for achieving appropriate analgesia following hip arthroscopy has not yet been defined. Determining means of achieving acceptable post-operative pain relief while minimizing narcotic usage will help yield maximal patient outcomes.The primary research procedures entailed in this study include fascia iliaca nerve blockade with Marcaine and local field infiltration with liposomal bupivicane (Exparel). The patients in this study will include those who have both a clinical and radiographic diagnosis of femoracetabular impingement (FAI), have failed non operative treatment, and are indicated for hip arthroscopy with labral repair and femoroplasty/acetabuloplasty. The study includes the surgical procedure and the first post-operative follow up visit. The total study duration is approximately 1.5 weeks for each patient. The study will be carried out until the patients first post-operative visit which typically occurs 7-10 days after the procedure. We are to include approximately 40 patients in total for this study over a period of 4 months.

ELIGIBILITY:
Inclusion Criteria:

* adult patients (>18 years old)
* diagnosed FAI that are indicated for hip arthroscopic labral repair and femoroplasty/acetabuloplasty.

Exclusion Criteria:

* patients undergoing revision procedures, bilateral procedures,
* advanced osteoarthritis (<2mm joint space on plain radiographs)
* frank dysplasia (anterior and/or lateral center edge angles <20 degrees and/or Tonnis angle >15 degrees)
* diagnoses other than FAI (Legg Calve Perthes, femoral head avascular necrosis, septic arthritis, or post traumatic deformity).
* allergy to liposomal bupivicaine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2019-10-29 (Actual); Primary Completion 2020-03-17 (Actual); Study Completion 2020-03-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Banffy, MD, Principal Investigator — Cedars Sinai
Locations (1):
- Kerlan Jobe, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mont MA, Beaver WB, Dysart SH, Barrington JW, Del Gaizo DJ. Local Infiltration Analgesia With Liposomal Bupivacaine Improves Pain Scores and Reduces Opioid Use After Total Knee Arthroplasty: Results of a Randomized Controlled Trial. J Arthroplasty. 2018 Jan;33(1):90-96. doi: 10.1016/j.arth.2017.07.024. Epub 2017 Jul 25. PMID 28802777
- [Background] Krych AJ, Baran S, Kuzma SA, Smith HM, Johnson RL, Levy BA. Utility of multimodal analgesia with fascia iliaca blockade for acute pain management following hip arthroscopy. Knee Surg Sports Traumatol Arthrosc. 2014 Apr;22(4):843-7. doi: 10.1007/s00167-013-2665-y. Epub 2013 Sep 24. PMID 24061718

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Liposomal Bupivicaine | Fascia Iliaca Blockade
Started | 20 | 17
Completed | 20 | 17
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Liposomal Bupivicaine | Fascia Iliaca Blockade | Total
Number analyzed (Participants) | 20 | 17 | 37
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 17 | 37
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 9 | 18
  Male | 11 | 8 | 19
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 20 | 17 | 37
BMI [Mean (Full Range); unit: Kg/m^2] — BMI utilized for each hip scope .It is a demographic characteristic not a result of the research medication that was being tested . As such, this as not analyzed and standard deviation is not necessary.
  Kg/m^2 | 26.4 [14 to 40] | 25.7 [14 to 40] | 26.05 [14 to 40]
Traction time [Mean (Full Range); unit: MINUTES] — Traction time s utilized for each hip scope .It is a demographic characteristic not a result of the research medication that was being tested . As such, this as not analyzed and standard deviation is not necessary.
  MINUTES | 36.0 [0 to 120] | 36.8 [0 to 120] | 36.4 [0 to 120]
pre-op Visual analogue scale score [Mean (Full Range); unit: CM] — Visual analogue scales (VAS) are psychometric measuring instruments designed to document the characteristics of disease-related symptom severity in individual patients and use this to achieve a rapid (statistically measurable and reproducible) classification of symptom severity and disease control. 0 equals no pain and 10 represents the worst pain.
  CM | 3.2 [0 to 10] | 2.2 [0 to 10] | 2.7 [0 to 10]

OUTCOME MEASURES:

1. Primary Outcome: Visual Analogue Scale
Description: pain scale Questionnaire 0 equals no pain at all and 10 equals the worst. The out come measure time frame is reported as the average VAS score of the first 4 day post op.
Time Frame: post op days 1-4 (Average VAS score of first 4 days of post op)
Measure: Mean (Full Range); unit: cm
Arm/Group | Liposomal Bupivicaine | Fascia Iliaca Blockade
Number analyzed (Participants) | 20 | 17
cm | 2.4 [1.5 to 3.8] | 2.7 [0.8 to 3.3]

2. Secondary Outcome: Narcotic Utilization
Description: Record of number of narcotic pain pills utilized by patients . This was reported as a total from post op day 1 to 4. The number listed is an average from each patient, from the total pills taken at home.
Time Frame: total pill taken over the course of days 1-4 post op.
Measure: Mean (Full Range); unit: number of pills
Arm/Group | Liposomal Bupivicaine | Fascia Iliaca Blockade
Number analyzed (Participants) | 20 | 17
number of pills | 7.6 [0 to 12] | 7.8 [0 to 12]

3. Secondary Outcome: Total Number of at Home Falls.
Description: number of falls occurring at home after discharge. This is the total number of falls of all patients in each group, over the first 7 days post op. This is not reported as a mean.
Time Frame: Post op days 1-7
Measure: Number; unit: total number of falls
Arm/Group | Liposomal Bupivicaine | Fascia Iliaca Blockade
Number analyzed (Participants) | 20 | 17
total number of falls | 0 | 6

ADVERSE EVENTS:
Time Frame: The adverse events occurred through post op days 1-7 for each patient.
Description: An adverse event is defined as a fall post op.
Arm/Group | Liposomal Bupivicaine | Fascia Iliaca Blockade
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/17
Other Adverse Events (participants affected / at risk) | 0/20 | 6/17
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Liposomal Bupivicaine (N=20) | Fascia Iliaca Blockade (N=17)
fall (Musculoskeletal and connective tissue disorders) | 0 (0) | 6 (6)

LIMITATIONS AND CAVEATS:
We did not meet target enrollment due to safety concerns.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-27): https://cdn.clinicaltrials.gov/large-docs/58/NCT04114058/Prot_SAP_002.pdf